CLINICAL TRIAL: NCT06769555
Title: A Single-arm Multi-center Trial of BCMA/CD3 Bispecific Antibody for Relapsed/Refractory AL Amyloidosis or Newly Diagnosed AL Amyloidosis With Insufficient Depth of Hematologic Response After Induction Therapy
Brief Title: BCMA/CD3 BiTE for RRAL or NDAL Amyloidosis With Insufficient Depth of Hematologic Response After Induction Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024012
Record Dates: First submitted 2024-12-10; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-06

CONDITIONS: AL Amyloidosis
Keywords: AL Amyloidosis; BCMA/CD3 BiTE; CM-336
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Intervention Model Description: A single-arm multi-center trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCMA/CD3 BiTE (Experimental)
  Interventions: Drug: CM-336 BCMA/CD3 bispecific antibody

INTERVENTIONS:
Drug: CM-336 BCMA/CD3 bispecific antibody — Patients received subcutaneous CM-336 80 mg once weekly in 28-d cycles after two step-up priming doses of 3 mg and 20 mg given on day 1 and day 4 of cycle 1. For patients achieve hematological PR or better after 2 cycles, and hematological VGPR or better after 4 cycles, the treatment regimen will change to 160mg once every 2 weeks (Q2W).

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness and safety of CM-336, which is a BCMA/CD3 BiTE, in patients with relapsed/refractory AL amyloidosis or newly diagnosed AL amyloidosis with insufficient depth of hematologic response after induction therapy.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate the effectiveness and safety of CM-336, which is a BCMA/CD3 BiTE, in patients with relapsed/refractory AL amyloidosis or newly diagnosed AL amyloidosis with insufficient depth of hematologic response after induction therapy.

Patients received subcutaneous CM-336 80 mg once weekly in 28-d cycles after two step-up priming doses of 3 mg and 20 mg given on day 1 and day 4 of cycle 1. For patients achieve hematological PR or better after 2 cycles, and hematological VGPR or better after 4 cycles, the treatment regimen will change to 160mg once every 2 weeks (Q2W).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years or older
* Biopsy-proven diagnosis of AL amyloidosis, according to the following standard criteria:
* Histochemical diagnosis of amyloidosis, as based on tissue specimens with Congo red staining with exhibition of an apple-green birefringence
* If clinical and laboratory parameters are insufficient to establish AL amyloidosis, or in cases of doubt, amyloid typing may be necessary
* Provide informed consent form
* Measurable disease, as defined by serum differential free light-chain concentration (dFLC; defined as the difference between amyloid forming [involved] and nonamyloid forming [uninvolved] free light-chain [FLC]) ≥50 mg/L)
* Received at least one prior line of therapy
* Must have been exposed to CD38 mAb
* Relapsed/refractory AL amyloidosis or newly diagnosed AL amyloidosis with insufficient depth of hematologic response after induction therapy
* Relapsed is defined as documented progressive disease >60 days after the last dose of prior therapy
* Refractory is defined as the documented absence of a hematologic response or hematologic progression on or within 60 days after the last dose of prior therapy
* Insufficient depth of hematologic response is defined as less than hematological PR by 2 cycles or less than hematologic VGPR by 4 cycles
* Eastern Cooperative Oncology Group performance status ≤3
* Clinical laboratory values:
* Absolute neutrophil count ≥1000/µL
* Platelet count ≥75,000/µL
* Hemoglobin ≥75g/L
* Total bilirubin ≤1.5× the upper limit of normal (ULN), except for patients with Gilbert's syndrome (as defined by >80% unconjugated bilirubin and total bilirubin ≤6 mg/dL)
* Alkaline phosphatase ≤5× ULN
* Alanine aminotransferase or aspartate aminotransferase ≤3× ULN
* Calculated creatinine clearance ≥30 mL/min
* The woman is not breastfeeding, is not pregnant, and agrees not to be pregnant during the study period and for the following 12 months.
* Male patients agreed that their spouse would not become pregnant during the study period and for 12 months thereafter.

Exclusion Criteria:

* Non-AL amyloidosis, including hereditary amyloidosis
* Diagnosed with multiple myeloma, according to the International Myeloma Working Group criteria
* Have been exposed to BCMA-targeted treatment
* Known intolerance, hypersensitivity, or contraindication to BCMA BiTE cellular products
* Patients with peripheral neuropathy greater than grade 2 or peripheral neuropathy greater than grade 2 with pain at baseline, regardless of whether they were currently receiving medical therapy, after excluding AL amyloidosis-related peripheral neuropathy
* Medically documented cardiac syncope, myocardial infarction within the previous 6 months, unstable angina pectoris, clinically significant repetitive ventricular arrhythmias despite antiarrhythmic treatment, or severe orthostatic hypotension or clinically important autonomic disease
* Ongoing or active infection, known HIV-positive status, or active hepatitis B or C infection
* Women who are pregnant or breastfeeding
* Subjects had major surgery within 2 weeks before randomization (for example, general anesthesia), or have not fully recovered from the surgery, or surgery is arranged during the study period
* Received live attenuated vaccine within 4 weeks prior to study treatment
* According to the researcher's judgment, any condition including but not limited to serious mental illness, medical illness, or other symptoms/conditions that may affect study treatment, compliance, or the capability of providing informed consent.

Necessary medication or supportive therapy is contraindicated with study treatment.

Any diseases or complications that may interfere with the study. Patients are not willing to or cannot comply with study scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Hematologic response VGPR or better rate after four cycles | Four months
  Hematologic response VGPR or better rate based on central laboratory results and the 2010 International Society of Amyloidosis (ISA) Consensus Criteria as evaluated by an Adjudication Committee (AC)
Adverse events and serious adverse events | Up to 2 year
  Adverse events (AEs), serious adverse events (SAEs), according to Common Terminology Criteria for Adverse Events (CTCAE) 5.0

SECONDARY OUTCOMES:
Time to hematologic response | Up to 2 year
  Time from randomization to first documentation of hematologic response
Hematologic best response | Up to 2 year
  Best Hematologic response allowed at study entry according to central laboratory results and International Society of Amyloidosis criteria as evaluated by an AC
Duration of hematologic response | Up to 2 year
  Time from the date of first documentation of hematologic response to the date of first documented hematologic disease progression, respectively according to central laboratory results and ISA criteria as determined by an AC
Hematologic response rate | Up to 2 year
  Overall hematologic (CR + VGPR + PR) response rate based on central laboratory results and the 2010 International Society of Amyloidosis (ISA) Consensus Criteria as evaluated by an AC
Overall survival | Up to 5 year
  Time from randomization to date of death. Patients without documentation of death at the time of analysis were censored at the date last known to be alive
Progression-free survival | Up to 5 year
  Time from randomization to date of hematologic progression. Patients without documentation of death at the time of analysis were censored at the date last known to be alive
Vital organ best response | Up to 2 year
  Best response in the vital organs allowed at study entry (heart and kidney) according to central laboratory results and International Society of Amyloidosis criteria as evaluated by an AC
Vital organ progression-free survival | Up to 2 year
  Time from randomization to first documentation of vital organ (heart or kidney) progression* or death due to any cause, whichever occurred first. Patients without documentation of vital organ (heart or kidney) progression* were censored at the date of last organ assessment of stable disease or better

IPD SHARING:
Plan to Share IPD: No